CLINICAL TRIAL: NCT03626441
Title: An Evaluation of the Effectiveness of a Single Dose of Preoperative Ginger on the Incidence of Postoperative Nausea and Vomiting in Patients Undergoing Elective Gynaecological Surgery
Brief Title: The Effect of Ginger on the Incidence of Postoperative Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Patrick J Toppin, Associate lecturer, The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Anaesthesia20182
Record Dates: First submitted 2018-07-14; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative Nausea and Vomiting; Ginger
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — ginger extract

STUDY DESIGN:
Intervention Model Description: Quadruple, blind randomized, controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sequentially numbered, sealed, opaque envelopes prepared and opened the evening before the surgery. Tablets containing either placebo or ginger allocated by a person not involved in any other aspect of the study and administered on the morning of surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Two coloured capsules containing 0.5 mg of cornstarch and flavoured with non-active essence of ginger, given 2 hours before the scheduled start of surgery.
  Interventions: Dietary Supplement: Placebo
- Ginger (Experimental): Two coloured capsules containing 0.5g ginger powder, flavoured with non-active essence of ginger, given 2 hours before the scheduled start of surgery.
  Interventions: Dietary Supplement: Ginger; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ginger — Capsules containing 0.5g ginger powder, flavoured with non-active essence of ginger
  Arms: Ginger
Dietary Supplement: Placebo — Two coloured capsules containing 0.5 mg of cornstarch and flavoured with non-active essence of ginger.

SUMMARY:
This study evaluates the effectiveness of ginger on the incidence of postoperative nausea and vomiting in patients undergoing gynaecological surgery. Half the patients were given an oral dose of ginger preoperatively and half received placebo.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) commonly complicate surgery and may lead to a prolonged length of stay in hospital, increased complication rates and decreased patient satisfaction. Gynaecological surgery is considered high risk for PONV.

Ginger is a cheap, widely available and safe natural product in Jamaica and has been found to reduce the incidence of Nausea and vomiting in other clinical situations, such as in pregnancy. It is believed to act via the inhibition of serotonergic receptors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Undergoing elective intra-abdominal, gynaecological surgery

Exclusion Criteria:

* Allergy to ginger, ginger by-products or cornstarch
* Gastroesophageal reflux disease (GERD)
* Allergy to any of the Anaesthesia Agents
* Inability to swallow capsules.
* psychiatric illness which prevents patients giving informed consent.
* Psychological which prevents patients giving informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-12-02 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
Incidence of post operative nausea or vomiting | 12 hours after surgery
  The proportion of patient who have any episodes of nausea or vomiting following surgery

SECONDARY OUTCOMES:
Severity of post operative Nausea and vomiting | 12 hours after surgery
  Measured using the Rhodes index
Severity of post operative Nausea and vomiting | 24 hours after surgery
  Measured using the Rhodes index
Severity of post operative Nausea and vomiting | 48 hours after surgery
  Measured using the Rhodes index
Severity of post operative Nausea and vomiting | 12 hours after surgery
  Measured using the BARF scale
Severity of post operative Nausea and vomiting | 24 hours after surgery
  Measured using the BARF scale
Severity of post operative Nausea and vomiting | 48 hours after surgery
  Measured using the BARF scale
Patient satisfaction | 48 hours post surgery
  Measured using a questionnaire administered to patient by investigators

CONTACTS AND LOCATIONS:
Overall Officials: Hyacinth Harding, DM, Principal Investigator — UWI, Faculty of medical sciencces; Andrea Myers, MD, Study Director — UWI, Faculty of medical sciencces
Locations (1):
- University of the West Indies, Kingston, Kng 7, Jamaica

IPD SHARING:
Plan to Share IPD: No
There is no plan to make patient data available to other researchers